CLINICAL TRIAL: NCT05428995
Title: A Randomized Comparison Between the C-MAC and Airtraq Videolaryngoscopes for First-attempt Intubation Success in Awake Patients With Anticipated Difficult Airway.
Brief Title: Comparison of Two Videolaryngoscopes (C-MAC vs Airtraq) for Awake Intubation
Acronym: AWAKECMACTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Manuel Taboada Muñiz, Professor University Of Santiago de Compostela, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AWAKE-CMAC-AIRTRAQ
Record Dates: First submitted 2022-06-15; First posted 2022-06-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-07

CONDITIONS: Intubation
Keywords: intubation; difficult airway; videolaryngoscope

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-MAC videolaryngoscope (Active Comparator): Patients with anticipated difficult airway will be awake intubated with a C-MAC videolaryngoscopy. Spontaneous breathing will be preserved, and the same protocol of sedation plus upper airways topical anesthesia will be applied in both groups.
  Interventions: Device: C-MAC videolaryngoscope
- Airtraq videolaryngoscope (Active Comparator): Patients with anticipated difficult airway will be awake intubated with a Airtraq videolaryngoscopy. Spontaneous breathing will be preserved, and the same protocol of sedation plus upper airways topical anesthesia will be applied in both groups.
  Interventions: Device: Airtraq videolaryngoscope.

INTERVENTIONS:
Device: C-MAC videolaryngoscope — Patients with anticipated difficult airway will be awake intubated with a C-MAC videolaryngoscopy
  Arms: C-MAC videolaryngoscope
Device: Airtraq videolaryngoscope. — Patients with anticipated difficult airway will be awake intubated with a Airtraq videolaryngoscopy
  Arms: Airtraq videolaryngoscope

SUMMARY:
Patients with anticipated difficult airway are recommended to be managed with an awake tracheal intubation. Initially fibreoptic bronchoscopy was considered the gold standard, but in the last decade videolaryngoscopes have been demonstrated to be an efficacy alternative technique. Recently, a systematic review and meta-analysis was published investigating the efficacy and safety of videolaryngoscopy compared with fibreoptic bronchoscopy for awake tracheal intubation. Eight prospective, randomized studies were included, with different videolaryngoscopes (C-MAC, GlideScope, Pentax AWS, McGraft, and Bullard). However, a direct comparison of two different videolaryngoscopes for awake tracheal intubation in patients with anticipated difficult airway has not been performed.

DETAILED DESCRIPTION:
This is a clinical prospective randomized-controlled trial. The aim of this study is to compare two different devices (C-MAC videolaryngoscope and Airtraq videolaryngoscope) for awake tracheal intubation in patients with difficult airways scheduled for surgery. The primary endpoint will be to compare first-attempt intubation success rate between the two videolaryngoscopes. Secondary outcomes will be to compare: difference in the overall success rate, number of intubation attempts, Cormack-Lehane grade of glottic view, incidence of complications related to intubation, difficulty experienced by the operator, patient's tolerability of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patients with anticipated difficult airway requiring awake intubation under local anaesthesia and conscious sedation for general anesthesia.
* Written informed consent from the patient or proxy (if present) before inclusion or once possible when patient has been included in a context of emergency.

Exclusion Criteria:

* Pregnancy
* age <18 years
* refusal of the patient
* patient's respiratory failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Difference in the first attempt intubation success rate (percentage) | during intubation
  To compare the difference in the first attempt success rate (percentage) of different awake videolaryngoscope techniques for tracheal intubation.

SECONDARY OUTCOMES:
Difference in the overall success rate (percentage) | during intubation
  To compare the difference overall success rate (percentage) with the two awake videolaryngoscope techniques for tracheal intubation.
Number of intubation attempts | during intubation
  To compare number of intubations attempts with the two awake videolaryngoscope techniques.
Cormack-Lehane grade of glottic view | during intubation
  To compare Cormack-Lehane grade of glottic view with the two awake videolaryngoscope techniques for tracheal intubation.
Difference in the incidence of complications related to intubation (percentage) | Participants will be followed from the beginning of the intervention to 30 minutes after the intervention
  To compare the difference in complications (percentage) with the two awake videolaryngoscope techniques. Hypoxemia (SpO2) < 90 %, Hypoxemia severe (SpO2) < 80 %, Hypotension defined as systolic blood pressure less than 80 mm Hg Severe hypotension defined as systolic blood pressure less than 65 mm Hg Cardiac arrest, death during intubation Moderate or difficult intubation esophageal intubation pulmonary aspiration, dental injuries Oral-pharynx and larynx traumatism
Degree of subjective difficulty experienced by the operator | during intubation
  Operator-assessed subjective difficulty of intubation by means of a special analogue numerical scale from 0 to 10, where 0=no subjective difficulty and 10=maximal subjective difficulty
Degree of subjective patient's tolerability of the procedure | during intubation
  Operator-assessed subjective patient's tolerance of the procedure by means of a special analogue numerical scale from 0 to 10, where 0=very good subjective tolerance and 10=very bad subjective tolerance
Degree of patient's confort of the procedure | 24 hours after intubation
  During the postoperative visit on the following day (24 hours after intubation), patient will be asked to rate their confort during the procedure by means of a special analogue numerical scale from 0 to 10, where 0=very good tolerance and 10=worst possible discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Taboada Muñiz, Ph.D., Principal Investigator — University Clinical Hospital of Santiago de Compostela
Locations (1):
- University Clinical Hospital of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data How to access data: Requests must be sent to manutabo@yahoo.es When available: With publication Additional Information Who can access the data: Researchers whose proposed use of the data has been approved Types of analyses: For scientific purpose Mechanisms of data availability: With investigator support
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When available: With publication
Access Criteria: Researchers whose proposed use of the data has been approved Types of analyses: For scientific purpose

REFERENCES:
- [Background] Alhomary M, Ramadan E, Curran E, Walsh SR. Videolaryngoscopy vs. fibreoptic bronchoscopy for awake tracheal intubation: a systematic review and meta-analysis. Anaesthesia. 2018 Sep;73(9):1151-1161. doi: 10.1111/anae.14299. Epub 2018 Apr 17. PMID 29687891
- [Background] Lewis SR, Butler AR, Parker J, Cook TM, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adult patients requiring tracheal intubation. Cochrane Database Syst Rev. 2016 Nov 15;11(11):CD011136. doi: 10.1002/14651858.CD011136.pub2. PMID 27844477
- [Background] Moore A, Schricker T. Awake videolaryngoscopy versus fiberoptic bronchoscopy. Curr Opin Anaesthesiol. 2019 Dec;32(6):764-768. doi: 10.1097/ACO.0000000000000771. PMID 31356364
- [Background] Moore AR, Schricker T, Court O. Awake videolaryngoscopy-assisted tracheal intubation of the morbidly obese. Anaesthesia. 2012 Mar;67(3):232-5. doi: 10.1111/j.1365-2044.2011.06979.x. PMID 22321077